CLINICAL TRIAL: NCT03166111
Title: Effect of Self-administered Lidocaine In-situ Gel Prior to Intrauterine Device Insertion in Women With no Previous Vaginal Delivery: A Randomized Controlled Study
Brief Title: Lidocaine In-situ Gel Prior to Intrauterine Device Insertion in Women With no Previous Vaginal Delivery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LISITU
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Contraception

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine group (Experimental): lidocaine in-situ gel inserted vaginally
  Interventions: Drug: lidocaine gel
- placebo group (Placebo Comparator): placebo gel inserted vaginally
  Interventions: Drug: placebo gel

INTERVENTIONS:
Drug: lidocaine gel — syringe filled with 5 ml gel to be self-administered vaginal 10 minutes prior to insertion
  Arms: lidocaine group
Drug: placebo gel — syringe filled with 5 ml gel to be self-administered vaginal 10 minutes prior to insertion
  Arms: placebo group

SUMMARY:
Long-acting reversible contraception methods are highly effective methods for reduction of the unplanned pregnancy rate worldwide. The intrauterine device is a single procedure that provides reliable, effective and long term contraception for many women. However, the insertion procedure can be associated with a troublesome degree of pain that prevent some women from choosing its use. Different interventions have been described to decrease pain perception during intrauterine device insertion with no agreement on an effective one. Pre-insertion oral ibuprofen, diclofenac, nitroprusside, local anesthetics as lidocaine and prostaglandins has been reported with variable degrees of success .

ELIGIBILITY:
Inclusion criteria:

* Non-pregnant women
* Women that did not receive any analgesics or misoprostol in the 24 hours prior to insertion
* Women who delivered only by caesarean section

Exclusion criteria:

* Women with any uterine abnormalities as congenital anomalies, endometrial lesions, adenomyosis, fibroids
* Those with a Category 3 or 4 conditions for intrauterine device insertion according to the WHO Medical Eligibility Criteria for contraceptive use
* Allergy to lidocaine.
* Women refuse to participate in the study

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
The difference in pain scores during intrauterine device insertion | 10 minutes
  using visual analog scale from 0 to 10

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abbas AM, Abd Ellah NH, Hosny MA, Abdellah MS, Ali MK. Self-administrated vaginal 2% lidocaine in-situ gel for pain relief during copper intrauterine device insertion in women with previous caesarean delivery only: a randomised, double-blind placebo-controlled trial. Eur J Contracept Reprod Health Care. 2021 Apr;26(2):132-138. doi: 10.1080/13625187.2020.1868427. Epub 2021 Feb 4. PMID 33539256